CLINICAL TRIAL: NCT03729271
Title: The Role of Breath Testing in Enriching the Likelihood of Response to Rifaximin in Patients With Diarrhea IBS
Brief Title: Hydrogen Breath Test an Instrument to Predict Rifaximin-Response in Irritable Bowel Syndrome Predominant Diarrhea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Commonwealth Diagnostics International, Inc. (Unknown)
Responsible Party: Principal Investigator, William Chey, Professor of Internal Medicine, Medical School and Professor of Nutritional Sciences, School of Public Health, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00142925
Record Dates: First submitted 2018-10-10; First posted 2018-11-02 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-02

CONDITIONS: Irritable Bowel Syndrome; Irritable Bowel Syndrome With Diarrhea
Keywords: IBS; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Rifaximin

STUDY DESIGN:
Masking Description: The study drug will be open label. However, the order of the breath tests that are performed (glucose and lactulose) will be blinded to the participant and the person performing the breath sample, and the results of the breath test.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Rifaximin and breath tests (Experimental): Rifaximin 550mg three times a day for 14 days. Breath tests (glucose and lactulose) will be completed prior to Rifaximin treatment and at week 13 of the study.
  Interventions: Drug: Rifaximin; Device: Glucose and lactulose hydrogen breath testing

INTERVENTIONS:
Drug: Rifaximin — Rifaximin will be given during weeks 2-4
  Other Names: Xifaxan
Device: Glucose and lactulose hydrogen breath testing — Subjects will undergo glucose and lactulose hydrogen breath tests for Small Intestinal Bacterial Overgrowth (SIBO) on consecutive days using a commercially available home base kits (Glucose Hydrogen Breath Test Collection Kit and Lactulose Hydrogen Breath Test Collection Kit for SIBO from Commonwealth Diagnostic International) prior to Rifaximin treatment and at week 13 of the study.

SUMMARY:
The purpose of this study is to learn more about how to improve treatment of patients with diarrhea predominant Irritable Bowel Syndrome (IBS-D) symptoms.Included patients will be requested to answer online surveys and will undergo treatment with rifaximin. Hydrogen breath testing and biologic samples collection will also be completed during the study.

DETAILED DESCRIPTION:
The study aims to determine whether hydrogen breath testing can be used to identify patients with IBS-D who are more likely to respond to rifaximin. Participating patients will complete a one week screening period when brief daily survey will be answered. Eligible patients will proceed with the treatment phase of the study, when patients will receive a 14 day course of rifaximin. All included patients will complete glucose and lactulose hydrogen breath tests before and after rifaximin treatment. Biological samples (e.g. blood, stool) will be collected at pre-determined time points and patients will answer daily brief survey for the duration of the study.

It is anticipated that 210 patients will be screened to reach a goal of enrolling 175 patients for the treatment phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* IBS-D (Rome IV Diagnostic Criteria)
* Diary compliance for at least 5 days and no rescue medications during baseline
* Appropriate levels of abdominal pain and diarrhea

Exclusion Criteria:

* Pregnant women or planning on becoming pregnant while in the study, or lactating women while in the study
* Inflammatory bowel disease, diabetes mellitus, systemic sclerosis, or celiac disease
* Active gastrointestinal or hematological malignancy which requires ongoing treatment
* Surgery to the GI tract in the past 3 months
* Gastrointestinal infection or diverticulitis in the past 3 months
* Severe hepatic impairment
* Any use of antibiotics in the past month
* Current use of probiotics
* Any history of allergies to rifaximin or its derivatives
* Any comitant use of P-glycoprotein inhibitors (for example. Cyclosporine)
* Known allergies to glucose or lactulose

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Number of treatment responders | first 4 weeks after rifaximin treatment
  A responder is defined as a patient simultaneously meeting weekly response criteria for abdominal pain (≥30% decrease from baseline in mean weekly pain score) and stool consistency (≥50% decrease from baseline in number of days/week with Bristol Stool Scale type 6 or 7 stool) during ≥2 of the 4 weeks after treatment

SECONDARY OUTCOMES:
Severity of abdominal pain by numeric rating scale (0-10) | baseline (week 1), up to 12 weeks
  A responder is defined as a patient with ≥30% decrease from baseline in mean weekly worst pain.
Stool consistency by Bristol Stool Form Scale (1-7) | baseline (week 1), up to 12 weeks
  A responder is defined as a patient with ≥ 50% decrease from baseline in number of days/weeks with Bristol stool scale type 6 or 7 stool.
Severity of bloating by numeric rating scale (0-10) | baseline (week 1), up to 12 weeks
  A responder is defined as a patient with ≥ 30 % decrease from baseline in mean weekly worst bloating score.
Severity of bowel urgency by rating scale (0-10) | baseline (week 1), up to 12 weeks
  A responder is defined as a patient with ≥ 30 % decrease from baseline in mean weekly worst urgency score.
Compare the predictive value of a pre-treatment glucose vs. lactulose hydrogen breath test for symptomatic response to rifaximin in IBS-D patients. | baseline (week 1), up to 12 weeks
  Irritable Bowel Syndrome- Severity Scoring system (IBS-SSS) responder decrease in score of >75 points compared to baseline. The scoring range is from 0% to 500% with decreasing points indicating improvements in symptoms. Scores will be compared week 1 to those collected on weeks 4, 8, and 12.
Irritable Bowel Syndrome - Quality of Life Measure responder | baseline (week 1), up to 12 weeks
  Defined as a decrease in score of 14 points from the baseline assessment. The score range is from 34 to 170, with decreasing in score indicating improvement in symptoms. Scores will be compared week 1 to those collected on weeks 4, 8, and 12.
Compare the predictive value of a pre-treatment glucose or lactulose hydrogen breath test | first 4 weeks after rifaximin treatment
  We will compare the proportion of patients meeting the primary response definition stratified by positive or negative glucose or lactulose breath test results

CONTACTS AND LOCATIONS:
Overall Officials: William Chey, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States